CLINICAL TRIAL: NCT03490019
Title: Treatment of Infantile and Juvenile Patients With Bardet-Biedl-Syndrome With Metformin. Evaluation of a Visual Improvement as a Side Effect of the Pediatric Treatment of Adipositas - a Prospective Pilot Study Without Control
Brief Title: Treatment of Bardet-Biedl-Syndrome With Metformin for Evaluation of a Possible Visual Improvement
Acronym: BBS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: unrealizable wishes of national authorities
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBS V1.0
Record Dates: First submitted 2018-03-19; First posted 2018-04-06 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-02

CONDITIONS: Bardet-Biedl Syndrome; Visual Impairment
MeSH Terms: conditions — Bardet-Biedl Syndrome; Vision Disorders | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Prospective pilot study without control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin Therapy (Experimental): Metformin therapy once daily for 24 weeks with a dose of 500, 850 or 1000 mg depending on body weight
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 500, 850 or 1000 mg depending on body weight once daily for 24 weeks

SUMMARY:
In this prospective pilot study without control group children and young adults (10-25 years old) diagnosed with Bardet-Biedl syndrome and treated with Metformin for their adipositas will be evaluated for a possible additional effect of Metformin on visual acuity.

DETAILED DESCRIPTION:
Within experiments with animals a positive effect of Metformin concerning the photo receptors was shown. Several patients of the university hospital Tübingen with Bardet-Biedl-Syndrome and Metformin therapy due to their adipositas reported a subjective improvement of the visual acuity which was confirmed by opthalmologic tests.

This will be checked in a prospective pilot study without control group including children and young adults (10-25 years old) diagnosed with Bardet-Biedl syndrome and treated with Metformin for their adipositas. Therefore a possible additional effect of Metformin on visual acuity will be evaluated under controlled conditions.

ELIGIBILITY:
Inclusion Criteria:

* clinically confirmed Bardet-Biedl-syndrome
* Visual acuity between 0.05 and 0.8
* Age >=10 year to <25 years
* Visual field III4e or V4e with diameter >=5°, if II4e not seen
* informed consent of patient and/or legal representative

Exclusion Criteria:

* Hypoglycaemia (<50mg/dl)
* Therapy with Metformin within the last three months
* Participation in another clinical trial
* pregnancy, lactation
* any contra indication concerning Metformin therapy
* Renal failure (creatinine clearance < 60ml/min)
* any acute disorder accompanied by clouding of consciousness
* acute or chronic disorders possible accompanied by tissue hypoxia
* Liver insufficiency, alcohol abuse
* not fluent in German language

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | Baseline to day 210
  Course of visual acuity according to appropriate table

SECONDARY OUTCOMES:
Number of letters read | Baseline to day 210
  Course visual acuity defined as number of letters read
Results of Static perimetry | Baseline to day 210
  Course of results of static perimetry given by measurement of light contrast sensitivity within at least 5 central points.
Results of Kinetic perimetry | Baseline to day 210
  Course of results of kinetic perimetry given by mapping the visual field sensitivity boundaries using Goldmann perimetry
Electroretinogram (ERG) dim-flash | Baseline to day 210
  Course of values of ERG dim-flash
Electroretinogram (ERG) standard flash | Baseline to day 210
  Course of values of ERG standard flash at 3 ods/m2
Electroretinogram (ERG) cone-single-flash | Baseline to day 210
  Course of values of ERG cone-single-flash at 30cd/m2
Electroretinogram (ERG) 30-Hz-Flicker | Baseline to day 210
  Course of values of ERG measured by 30-Hz-Flicker in all patients
Visual evoked potential (VEP) - amplitude | Baseline to day 210
  Course of results of measurement of VEP amplitude
Visual evoked potential (VEP) - latency time | Baseline to day 210
  Course of results of measurement of VEP latency time
FST | Baseline to day 210
  Full-Field-Stimulus Threshold
optical coherence tomography (OCT) | Baseline to day 210
  Course of central thickness of retina measured by OCT

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Billing, PD Dr. med., Principal Investigator — Universtitätsklinikum Tübingen

IPD SHARING:
Plan to Share IPD: Undecided